CLINICAL TRIAL: NCT03721939
Title: BEnefit of Arterial Preparation by LONGitudinal Scoring Before Paclitaxel Eluting Balloon Angioplasty of the Superficial Femoral and Popliteal Artery
Brief Title: BEnefit of Arterial Preparation by LONGitudinal Scoring
Acronym: BELONG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VentureMed Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BELONG Study
Record Dates: First submitted 2018-10-21; First posted 2018-10-26 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- FLEX Scoring Catheter plus DEB (Experimental): The target lesion is prepared by the FLEX Scoring Catheter® with a 30° rotation between each passage. Angioplasty is performed during 3 minutes with paclitaxel-coated balloon(s) (PCB), all along the target lesion.
  Interventions: Device: FLEX Scoring Catheter

INTERVENTIONS:
Device: FLEX Scoring Catheter — Vessel preparation with the FLEX Scoring Catheter® with a 30° rotation between each passage is performed, followed by a DEB angioplasty.

SUMMARY:
The purpose of the artery preparation concept is to perform regular longitudinal micro-incisions on the inner side of the artery ("scoring") and therefore promote a regular expansion of atheroma by balloon inflation.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18-year-old, with symptomatic lower extremity occlusive arterial disease
* Rutherford class of symptom 2 to 5
* Atheromatous ≥ 70 % stenosis or occlusion of SFA and/or PA
* Absence of > 50% residual stenosis of the run-in vessels at the end of procedure
* Presence of at least one patent (no ≥ 50 % stenosis) run-off tibial or fibular vessel to the foot at the end of procedure
* De novo or restenotic lesions, including in-stent restenosis
* Willingness to participate in the study and signature of informed consent

Exclusion Criteria:

* Renal failure with glomerular filtration rate (GFR) 30 ml/min or below, estimated by the Cockroft-Gault equation.
* Women who are pregnant, lactating, or planning to become pregnant during the duration of the study
* Recent artery thrombosis, at risk of distal embolization during percutaneous procedure
* Previous use of a PCB in the lesion during last 15 months
* Extremely calcified lesions, defined by calcification involving ³ 270° of the artery circumference over ³ 15 cm.
* Sub-intimal recanalization
* Tortuous contra-lateral femoral access with difficult cross-over
* Previous or planned surgery of the target lesion
* High risk of bleeding
* Contra-indication to dual antiplatelet therapy for one month, and/or to single antiplatelet therapy for 1 year
* Allergy to aspirin, clopidogrel or heparin
* Life expectancy less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2024-03-04 (Actual)

PRIMARY OUTCOMES:
Absence of clinically driven target lesion revascularization (CDTLR) at 12 months | 12 months
Occurrence of death from cardiovascular origin | 12 months
Occurrence of major amputation of target limb | 12 months

SECONDARY OUTCOMES:
Primary patency of the treated lesion (defined by PSVR ≤ 2.5 at duplex scan) | 3 and 12 months
Absence of CDTLR | 3 months
Absence of major amputation | 3 and 12 months
Change in ankle brachial index (ABI) | 3 and 12 months
Change in Rutherford class of symptom | 3 and 12 Months
Technical success of the scoring procedure | Average of 2 hours
Proportion of luminal gain | Average of 2 hours
Occurrence of dissection | Average of 2 hours
Proportion of stent implantation | Average of 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Periard, MD, Principal Investigator — Fribourg Cantonal Hospital
Locations (1):
- Hôpital Cantonal de Fribourg, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: No